CLINICAL TRIAL: NCT05825911
Title: Evaluation of Diagnostic Accuracy of MCG Scan in Suspected Coronary Artery Disease
Brief Title: Evaluation of Diagnostic Accuracy of MCG(Magnetocardiography) Scan in Suspected Coronary Artery Disease
Acronym: EDAM-CAD
Status: Recruiting | Type: Observational
Sponsor: AMCG (Industry)
Responsible Party: Sponsor
Other Study IDs: AMCG-CT01
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
Keywords: Magnetocardiography scan; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rest/Stress MCG scan — All patients enrolled and receiving standard screening tests for CAD will undergo rest/stress MCG scan before CAG.
Diagnostic Test: Rest MCG scan — This is an normal adult population with age-, and sex-matched control group. All participants enrolled will undergo rest MCG scan.

SUMMARY:
This multicenter clinical trial is designed to evaluate the diagnostic accuracy of MCG scan in detecting significant CAD compared to the reference standard CAG.

DETAILED DESCRIPTION:
This is multicenter, prospective, observational trial to evaluate the diagnostic accuracy of magnetocardiography(MCG) scan in detecting significant coronary artery disease(CAD) compared to the reference standard coronary arteriography(CAG). Chest pain patients scheduled for CAG will be offered to enroll in this clinical trial and provide informed consent to undergo with a rest/stress MCG scan prior to CAG. This MCG scan with a new 96 channel superconducting quantum interference device(SQUID) system is radiation-free, contactless and takes less than ten minutes to complete. Multiple studies have shown that the diagnostic accuracy of stress MCG scan is quite high in identifying patients with symptomatic CAD. Results will be interpreted and compared to the results of cardiac SPECT stress test, if available, and CAG. Participants will be followed up to 30 days via phone call or chart review. 30 day major adverse cardiac event(MACE) will be recorded and correlated with initial MCG scan results.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 years of age at the time of enrollment
* Patient presenting for CAG
* Consents to having an MCG scan study

Exclusion Criteria:

* Patients unable to fit into MCG scan device
* Patients with implanted cardiac pacemakers/defibrillators
* Atrial fibrillation with rapid ventricular response
* Patients with other sustained or incessant arrhythmias
* Presence clinical suspicious of any acute coronary syndrome

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. MAIN STUDY: This is an adult population at varying risk for CAD who will present at multicenter for cardiovascular screening with CAG.
  2. SUB-STUDY: This is an normal adult population with age-, and sex-matched control group.
Sampling Method: Non-Probability Sample
Enrollment: 908 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of MCG scan | 1 day
  Compare the diagnostic accuracy of stress MCG scan in detecting significant CAD compared to the current standard reference coronary angiogram(CAG) with statistical analysis including sensitivity, specificity.

SECONDARY OUTCOMES:
Positive predictive value(PPV), Negative predictive value(NPV), and diagnostic accuracy of MCG scan | 1 day
  Comparison with CAG will be performed for those having stress MCG scan test with statistical analysis including PPV, NPV, and diagnostic accuracy.

OTHER OUTCOMES:
Major adverse cardiac event after 30 days of CAG | 1 month
  The frequency and percentage of MACE collected 30 days after the end of the CAG and the types of events are presented. At this time, major adverse cardiovascular events (MACEs) to be collected include death due to cardiovascular disease (CV Death), myocardial infarction (Nonfatal MI), and ischemic cardiovascular events (Ischemic CV events).
Comparison of MCG scan with cardiac SPECT test | 1 day
  Comparison with cardiac SPECT test will be performed with statistical analysis including sensitivity and specificity.
Comparison of sensitivity and specificity between stress MCG scan and stress ECG test | 1 day
  Comparison of sensitivity and specificity between stress MCG scan and stress ECG test

CONTACTS AND LOCATIONS:
Overall Officials: Hoseong Lee Deputy general manager, Study Director — AMCG
Locations (2):
- South Korea (2):
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Eunpyeong-gu
  - Gachon University Gil Medical Center, Incheon, Namdong-gu

IPD SHARING:
Plan to Share IPD: No